CLINICAL TRIAL: NCT04773717
Title: The Effect of High Dose Parenteral Ascorbic Acid On Microcirculation In Sepsis. Randomized Double-Blind Placebo-Controlled Trial
Brief Title: The Effect of High Dose Parenteral Ascorbic Acid On Microcirculation In Sepsis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lithuanian University of Health Sciences (Other)
Responsible Party: Principal Investigator, Andrius Pranskunas, Professor, Lithuanian University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BE-2-5
Record Dates: First submitted 2021-02-21; First posted 2021-02-26 (Actual); Last update posted 2021-03-03 (Actual); Status verified 2021-02

CONDITIONS: Sepsis; Septic Shock
Keywords: Sepsis; Microcirculation; Ascorbic acid
MeSH Terms: conditions — Sepsis; Shock, Septic | interventions — Ascorbic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ascorbic acid (Experimental): Patients received a high dose of intravenous ascorbic acid in four equal parts daily for 96 hours.
  Images of sublingual microcirculation were obtained at a baseline, after 0.5, 6, 12, 24, 48, 72, and 96 hours.
  Interventions: Drug: Ascorbic acid
- Placebo (Placebo Comparator): Patients received placebo solution matching ascorbic acid solution as four equal parts daily for 96 hours. Images of sublingual microcirculation were obtained at a baseline, after 0.5, 6, 12, 24, 48, 72, and 96 hours.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ascorbic acid — 200mg/kg/24h in four equal parts
  Arms: Ascorbic acid
Drug: Placebo — The same regimen as ascorbic acid.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the effect of high-dose ascorbic acid on microcirculation in sepsis.

DETAILED DESCRIPTION:
Adult patients with septic shock were enrolled within 24 hours following admission to the Central Department of Intensive Care in Lithuanian University of Health Sciences Hospital Kaunas Clinics.

Participants were randomly assigned to a placebo or ascorbic acid group in a 1:1 ratio. They were resuscitated according to Surviving Sepsis Campaign Guidelines. Additionally, they received an intravenous infusion of ascorbic acid either placebo. The dose of ascorbic acid was 200mg/kg/24h divided into four equal parts for 96 hours. Sublingual microcirculatory measurements were obtained, using an incident dark field (IDF) device.

ELIGIBILITY:
Inclusion Criteria:

* Patients with sepsis or septic shock within the first 24 hours after ICU admission.

Exclusion Criteria:

* Age < 18 years,
* Pregnancy,
* Advanced malignancy,
* History of kidney stone, glucose-6-phosphate deficiency, hemochromatosis, or solid organ transplantation,
* Oral mucosal inflammation or injury or technical difficulties in obtaining sublingual images.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2021-01-31 (Actual)

PRIMARY OUTCOMES:
Microvascular flow index (MFI) | Baseline, after 0.5, 6, 12, 24, 48, 72 and 96 hours
  Changes in MFI
Proportion of perfused small vessels (PPV) | Baseline, after 0.5, 6, 12, 24, 48, 72 and 96 hours
  Changes in PPV

CONTACTS AND LOCATIONS:
Locations (1):
- Lithuanian University of Health Sciences Hospital Kaunas Clinics, Kaunas, Lithuania

REFERENCES:
- [Derived] Belousoviene E, Pranskuniene Z, Vaitkaitiene E, Pilvinis V, Pranskunas A. Effect of high-dose intravenous ascorbic acid on microcirculation and endothelial glycocalyx during sepsis and septic shock: a double-blind, randomized, placebo-controlled study. BMC Anesthesiol. 2023 Sep 12;23(1):309. doi: 10.1186/s12871-023-02265-z. PMID 37700249